CLINICAL TRIAL: NCT04133818
Title: Feasibility of a One-day-and-a-half Multidisciplinary Education and Exercise Therapy Program for Patients With Low Back Pain: a 3-month Retrospective Open Pilot Study
Brief Title: Feasibility of a One-day-and-a-half for Patients With Low Back Pain
Acronym: LC-ONE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: LC-ONE; APHP190887 (Other: APHP)
Record Dates: First submitted 2019-03-21; First posted 2019-10-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Subacute or Chronic Low Back Pain
Keywords: Multidisciplinary education and exercise therapy program.; Physical activity; Rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multidisciplinary program.: Patients with subacute or chronic LBP for whom first-line treatments had failed but for whom an intensive multidisciplinary rehabilitation program was not indicated.
  Interventions: Behavioral: Multidisciplinary education and exercise therapy program

INTERVENTIONS:
Behavioral: Multidisciplinary education and exercise therapy program — Multidisciplinary program: one and a half day of education and exercise therapy about low back pain :
  * Lectures and explanations about low back pain
  * Physical activity
  * Relaxation

SUMMARY:
The purpose of this study was to assess the feasibility of a one-day-and-a-half no intensive multidisciplinary education and exercise therapy program in the subgroup of patients with subacute or chronic LBP for whom first-line treatments had failed but for whom an intensive multidisciplinary rehabilitation program was not indicated.

DETAILED DESCRIPTION:
Retrospectively, data of patients between 18 and 60 years who had benefited in the PMR unit of Cochin' hospital of a one-day-and-a-half no intensive multidisciplinary education and exercise therapy program are collected.

This no intensive multidisciplinary education and exercise therapy program is proposed by the PMR unit of Cochin' hospital to all patients with a subacute or chronic low back pain for whom first-line treatments had failed but for whom an intensive multidisciplinary rehabilitation program is not indicated.

It is done in group of 4 to 6 people, performed by medical doctors with experience in the management of patients with low back pain, physiotherapists, occupational therapists, and psychologist.

Data regarding feasibility of this program were recorded with autoquestionnaires that patients had to fill in during the program and 3 months after.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* subacute or chronic non-specific LBP ≥ 6 weeks
* no indication for an intensive multidisciplinary rehabilitation program according to the senior physician, a specialist in physical medicine and rehabilitation and/or rheumatology with a strong experience in the care of patients with non-specific LBP
* currently working
* written consent

Exclusion Criteria:

* inability to speak or read French
* cognitive impairment
* current sick leave
* history of intensive multidisciplinary rehabilitation program for LBP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subacute or chronic LBP for whom first-line treatments had failed but for whom an intensive multidisciplinary rehabilitation program was not indicated and who had benefited in PMR unit of Cochin' hospital of a no intensive multidisciplinary rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | 3 months
  Acceptability of the program by the patients (evaluated by a visual analog scale (VAS) between 0 and 100 with 100 representing the best acceptability and 0 the lowest acceptability)

SECONDARY OUTCOMES:
Efficiency | 3 months
  Efficiency of the program to diminish pain (evaluated by a visual analog scale (VAS) between 0 and 100 with 100 representing the most important pain and 0 no pain at all)
Efficiency | 3 months
  Efficiency of the program to diminish fear and beliefs (FABQ, between 0 and 66 with 66 representing the highest level of fear and beliefs about low back pain and 0 representing no fear and beliefs about low back pain)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD, PhD, Principal Investigator — APHP (Assistance Publique-Hôpitaux de Paris)
Locations (1):
- Hôpital Cochin, Paris, France, France

REFERENCES:
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Adnan R, Van Oosterwijck J, Cagnie B, Dhondt E, Schouppe S, Van Akeleyen J, Logghe T, Danneels L. Determining Predictive Outcome Factors for a Multimodal Treatment Program in Low Back Pain Patients: A Retrospective Cohort Study. J Manipulative Physiol Ther. 2017 Nov-Dec;40(9):659-667. doi: 10.1016/j.jmpt.2017.09.001. PMID 29229056
- [Background] Brox JI, Storheim K, Grotle M, Tveito TH, Indahl A, Eriksen HR. Systematic review of back schools, brief education, and fear-avoidance training for chronic low back pain. Spine J. 2008 Nov-Dec;8(6):948-58. doi: 10.1016/j.spinee.2007.07.389. Epub 2007 Nov 19. PMID 18024224
- [Background] Garofoli R, Boisson M, Segretin F, Linieres J, Gerard C, Moreau S, Ieong E, Chagny F, Bedin C, Lefevre-Colau MM, Rannou F, Roren A, Nguyen C. Feasibility of a short multidisciplinary education and exercise therapy program for patients with non-specific low back pain: A 3-month retrospective open pilot study. Ann Phys Rehabil Med. 2019 Sep;62(5):382-385. doi: 10.1016/j.rehab.2019.05.005. Epub 2019 May 31. No abstract available. PMID 31158552